CLINICAL TRIAL: NCT03927261
Title: A Phase 1/1b Safety Study of PRGN-3006 Adoptive Cellular Therapy in Patients with CD33-Positive Relapsed or Refractory Acute Myeloid Leukemia, Minimal Residual Disease Positive Acute Myeloid Leukemia, and Higher Risk Myelodysplastic Syndrome
Brief Title: PRGN-3006 Adoptive Cellular Therapy for CD33-Positive Relapsed or Refractory AML, MRD Positive AML or Higher Risk MDS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Precigen, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRGN3006-001
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation and Dose Expansion of PRGN-3006 (Experimental): Participants will be treated in dose expansion phase to evaluate the safety and efficacy of the identified dose of PRGN-3006.
  Interventions: Drug: PRGN-3006 T Cells

INTERVENTIONS:
Drug: PRGN-3006 T Cells — Participants will receive up to 2 intravenous (IV) administrations of PRGN-3006 T Cells with or without lymphodepletion and will be monitored for safety, efficacy, and correlative endpoints for up to 12 months following infusion.

SUMMARY:
This is a first-in-human dose escalation/dose expansion study to evaluate the safety and identify the best dose of modified immune cells, PRGN-3006 (autologous chimeric antigen receptor (CAR) T cells), in adult patients with relapsed or refractory acute myeloid leukemia (AML), Minimal Residual Disease (MRD) positive acute myeloid leukemia or higher risk myelodysplastic syndrome (MDS). Autologous CAR T cells are modified immune cells that have been engineered in the laboratory to specifically target a protein found on tumor cells and kill them.

DETAILED DESCRIPTION:
This is a multi-center, nonrandomized, Phase 1/1b safety and tolerability study. The safety and tolerability of PRGN-3006 T cells will be assessed following intravenous administration of escalating doses in patients with relapsed or refractory CD33-positive AML, MRD-positive AML, or higher risk MDS.

This study has completed the dose escalation phase and is further evaluating PRGN-3006 at the identified dose in the dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with either relapsed or refractory AML (including extramedullary disease), MRD-positive AML, or higher risk MDS.
* Absolute lymphocyte count ≥ 0.2 k/μL.
* Karnofsky performance status score ≥60%.
* Life expectancy ≥ 12 weeks from the time of enrollment.
* Pretreatment calculated or measured creatinine clearance (absolute value) of ≥ 40 mL/minute or Cr < 2x upper limit of normal (ULN).
* Bilirubin ≤ 2.0 mg/dL or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in participants with well documented Gilbert's syndrome or hemolysis or who require regular blood transfusions
* Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) < 3.0 x ULN.
* Ejection fraction measured by echocardiogram (ECHO) or multi gated acquisition scan (MUGA) > 45%.
* Participant does not require supplemental oxygen or mechanical ventilation AND has an oxygen saturation by pulse oximetry of ≥ 92% or higher on room air.
* Negative serum pregnancy test. Note: Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for at least 1 year following study treatment (T cell infusion); should a woman participant or female partner of a male participant become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately.
* Participant has a matched bone marrow donor and is otherwise able to receive a bone marrow transplant (dose escalation phase only and for participants with MRD-positive AML)
* Participants who have undergone allo-SCT and/or donor lymphocyte infusion (DLI) are eligible if they are at least 3 months post SCT, prior to apheresis, atleast 30 days post last DLI prior to apheresis, have not received treatment or prophylaxis for GVHD 6 weeks before administration of CAR T cells, have no active GVHD.
* All participants must have the ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL M3): t(15;17)(q22;q12); (promyelocytic leukemia [PML]/retinoic acid receptor [RAR] alpha [a]) and variants excluded.
* Participants with peripheral blood blasts >35%
* Known central nervous system (CNS) leukemic involvement that is refractory to intrathecal chemotherapy and/or cranio-spinal radiation; participants with a history of CNS disease that have been effectively treated to complete remission ( i.e. no blasts in cerebrospinal fluid [CSF] by cytology and flow cytometry) will be eligible.
* Prior treatment with investigational CD33 targeting CAR T therapy for any disease.
* Prior treatment with licensed or investigational CD33 targeting monoclonal antibody or antibody drug conjugate within 6 months of apheresis.
* Participants enrolled in another investigational therapy protocol for their disease within 14 days or 5 half-lives of apheresis, whichever is shorter.
* Ongoing uncontrolled serious infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, poorly controlled pulmonary disease or psychiatric illness/social situations that would limit compliance with study requirements.
* Human immunodeficiency virus (HIV) seropositivity, or active hepatitis B or C infection based on testing performed within 28 days of enrollment.
* Participants requiring agents other than hydroxyurea to control blast counts within 14 days of study enrollment.
* Participants with presence of other active malignancy within 1 year of study entry; participants with adequately resected basal or squamous cell carcinoma of the skin, or adequately resected carcinoma in situ (e.g. cervix) may enroll irrespective of the time of diagnosis.
* Pregnant and lactating women are excluded from this study
* History of allergic reactions attributed to compounds of similar chemical or biological composition to cetuximab (anti-EGFR).
* Active autoimmune disease requiring systemic immunosuppressive therapy (i.e. >10mg of prednisone daily or equivalent).
* Participant, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience Dose Limiting Toxicities (DLTs) | Up to Day 42
  Incidence of dose limiting toxicity (DLT) as defined in the protocol
Number of Participants who Experience Treatment Emergent Adverse Events (TEAEs) | Up to 12 months post treatment
  Systemic toxicity in general and hematologic toxicity in specific will be assessed through the capture of TEAEs at each study visit and through laboratory assessments throughout the study. The severity of the TEAEs will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 scale.

SECONDARY OUTCOMES:
Disease Progression in AML Participants | Up to 12 months post treatment
  Proportion of AML patients achieving partial response (PR), complete response (CR), CR with incomplete count recovery (CRi), and/or morphologic leukemia free state (MLFS) by ELN Response Criteria in AML. CRh will also be captured, defined as <5% of blasts in the bone marrow, no evidence of disease, and partial recovery of peripheral blood counts.
Disease Response in MDS Patients | Up to 12 months post treatment
  Proportion of MDS patients achieving a response (CR, PR or Marrow CR) as defined in International Working Group (IWG) 2006 Criteria.
Rate of Absolute Neutrophil Count Recovery | Day 28
  Rate of Absolute Neutrophil count recovery (>0.5 x 10^9/L)
Absolute Lymphocyte Count (ALC) | Baseline
  ALC including CD4/CD8 subsets by flow cytometry at baseline (at apheresis) in patients who have successful versus failed PRGN-3006 production.
Number of PRGN-3006 T Cells | Up to 12 months post treatment
  Number of PRGN-3006 T Cells present in patients treated with PRGN-3006

CONTACTS AND LOCATIONS:
Overall Officials: Amy R. Lankford, PhD, Study Director — Precigen, Inc
Locations (2):
- United States (2):
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sallman DA, Elmariah H, Sweet K, Talati C, Mishra A, Cox CA, Semnani R, Shah RR, Sabzevari H, Chakaith M, Uthuppan J, Lankford A, Wang C, Padron E, Kuykendall AT, Komrokji RS, Lancet JE, Davila ML, Bejanyan N. Phase 1/1b Safety Study of Prgn-3006 Ultracar-T in Patients with Relapsed or Refractory CD33-Positive Acute Myeloid Leukemia and Higher Risk Myelodysplastic Syndromes. Blood. 2021; 138(Supplement 1):825.
- [Background] Sallman DA, Elmariah H, Sweet K, Mishra A, Cox CA, Chakaith M, Semnani R, Shehzad S, Anderson A, Sabzevari H, Lankford A, Chan O, SanchezMolina L, Wang C, Padron E, Kuykendall A, Komrokji RS, Lancet JE, Davila ML, Bejanyan N. Phase 1/1b Safety Study of Prgn-3006 Ultracar-T in Patients with Relapsed or Refractory CD33-Positive Acute Myeloid Leukemia and Higher Risk Myelodysplastic Syndromes. Blood. 2022; 140(Supplement 1):10313-10315.